CLINICAL TRIAL: NCT01440634
Title: Community-Based Detection and Treatment of Peripheral Arterial Disease in Hispanics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carlos H Timaran, Associate Professor of Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0830128N
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Community Medicine; Exercise Test; Exercise Therapy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- supervised exercise (Other): It consists of six months of supervised, intermittent track walking to near maximal leg pain or discomfort three days per week. Walking duration will begin at 20 - 30 minutes per session for the first month of the program, and increased by 5 minutes per session per month until a total of 45 minutes of walking per session is reached by the third month.
  Interventions: Other: Supervised exercise Program
- Standard of Care (No Intervention): Patients will be observed during the time of the study, no intervention will be applied. Patients are allowed to do their regular activity at home.

INTERVENTIONS:
Other: Supervised exercise Program — Supervised exercise Program consist of six months of supervised, intermittent track walking. Walking duration will begin at 20 - 30 minutes per session for the first month of the program, and increased by 5 minutes per session per month until a total of 45 minutes of walking per session is reached by the third month. During each exercise session, individuals will be encouraged to walk at a speed of approximately 2 mph until they achieve leg pain or discomfort on walking of moderate severity.Individuals are then allowed to have a brief period of standing or sitting rest to permit symptoms to resolve before they resume exercise.
  Arms: supervised exercise

SUMMARY:
Peripheral Arterial Disease (PAD) is a highly prevalent public health problem that results from progressive atherosclerosis of arteries in the lower extremities. PAD is also associated with major detrimental effects on quality of life and functional status, and is the most important cause of limb amputation. More importantly, PAD is a major manifestation of cardiovascular disease and a potent predictor of myocardial infarction, stroke and death. Despite its frequent occurrence, little is known about the natural history of PAD in Hispanics who represent 12.5% of the United States. Because access to health care is limited among Hispanics, CBPR is the ideal process to reach this target population. The goal of the proposed study is to evaluate community-based strategies of detection and treatment of peripheral arterial disease (PAD) in Hispanics. The proposed project consists of two phases: a cross-sectional phase (PAD detection), followed by a randomization phase.During the PAD detection study , the prevalence and severity of PAD in this population will be determined. Specific risk factors associated with PAD among the Hispanic participants will be identified. During the second phase patients will be enrolled in a randomized, non-blinded trial comparing a community-based risk factor modification and supervised exercise program versus usual care for PAD. These individuals will undergo a baseline evaluation similar to the one obtained during the first phase of the study, but will also include functional testing of the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

Cross-Sectional phase:

* Hispanic men and women aged 70 years or older.
* Hispanic participants with diabetes mellitus or smokers aged 50 through 69 years.
* Individual has been informed of the nature, procedures and risks of the study, and has signed a consent form approved by UT Southwestern Institutional Review Board.

Randomization phase:

* Hispanic men and women aged 70 years or older
* English or Spanish speaking
* Hispanic participants with diabetes mellitus or smokers aged 50 through 69 years.
* Documented peripheral arterial disease with an Ankle-brachial index (ABI) < 0.9 or Toe-brachial index (TBI) <0.7, and abnormal Pulse Volume Recordings (PVR).
* Ability to ambulate independently.
* No prior amputations other than toe or partial foot amputations that do not impede walking.
* Patient has been informed of the nature, procedures and risks of the study, and has signed a consent form approved by the UT Southwestern Institutional Review Board.

Exclusion Criteria:

Cross-Sectional Phase

* Individuals with severe dementia.
* Individuals with inability to provide informed consent.
* Bilateral lower or upper extremities amputations.
* Pregnancy or lactation. Randomization Phase
* Non-ambulatory
* Individuals with prior below- or above-knee amputations
* Individuals unable to give informed consent
* Individuals unwilling to perform the functional tests or quality of life assessments
* Individuals unable to perform exercise therapy, functional tests or quality of life assessments due to severe comorbidities
* Presence of concurrent illness with an anticipated life expectancy less than six months
* Individuals with planned operative interventions

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 347 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Timaran, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at community centers. Enrollment was performed between february 2008 and June 2011.
Pre-assignment Details: Patients that denied to be randomized and/or to follow the schedule for the research procedures was excluded of the study.
Period: Cross Sectional Phase
Arm/Group | Supervised Exercise | Standard of Care
Started | 0 | 347
Completed | 0 | 347
Not Completed | 0 | 0
Period: Randomization Phase
Arm/Group | Supervised Exercise | Standard of Care
Started | 30 | 24
Completed | 24 | 14
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supervised Exercise | Standard of Care | Total
Number analyzed (Participants) | 24 | 14 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 24 | 14 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75 [68 to 82] | 79.5 (11.08) [70.5 to 86] | 79.5 (11.08) [70.5 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Effect of an Exercise Intervention on Walking Ability (Functional Outcome)
Description: Walking distance (Six-Minute Walk test). Following a standardized protocol, individuals are instructed to walk back and forth a 100-ft hallway as far as they can in six minutes after instructions to cover as much distance as possible. A research assistant walks slightly behind each participant so as not to pace the individual. The research assistant records whether or not each person stops during the 6-minute walk. During the proposed study, members of the research team and trained lay health promoters (LHPs) will walk directly behind the individuals and give standardized instructions of encouragement at set intervals. Data will be reported on meters walked.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supervised Exercise | Standard of Care
Number analyzed (Participants) | 30 | 24
meters | 301.4 (140.3) | 185.1 (164.1)

ADVERSE EVENTS:
Arm/Group | Supervised Exercise | Standard of Care
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/30 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supervised Exercise (N=30) | Standard of Care (N=24)
Death (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was limited by the lack of patients compliance to follow the schedule for the exercise sessions. Patients did not assisted regularly to the walking sessions, and the schedule was completed in 70 % of the plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No